CLINICAL TRIAL: NCT01682122
Title: Evaluation of the Frequency and Persistence of Wide Pulse Pressure in the Neonatal Population
Brief Title: Frequency and Persistence of Wide Pulse Pressure in the Neonatal Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Philip Roth, MD, PhD, Director of Neonatology Chairman, Dept. of Pediatrics, & Vice President of Medical Education, Staten Island University Hospital
Other Study IDs: SIUH12-037; SIUH12-037 (Other: Staten Island University Hospital - IRB)
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Blood Pressure; Pediatrics; Infant, Newborn; Cardiology
Keywords: Blood Pressure; Pediatrics; Infant, Newborn; Cardiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Newborns: Healthy newborns in Regular and Observation nurseries who are between 0-72 hrs of age. Infants with gestational age > or = 35weeks and birth weight > 2500g, who are hemodynamically stable, have no cardiorespiratory abnormalities and have no evidence of sepsis. If a blood culture was drawn due to the presence of maternal risk factors (e.g. maternal fever, prolonged rupture of membranes), patients will be included only if the blood culture result is negative and in case of intrapartum antibiotic treatment, ancillary blood tests (CBC with differential, CRP) are also within the normal range

SUMMARY:
Wide Pulse Pressure is frequently present in the normal, full-term neonatal population. This study will evaluate the frequency and persistence of wide pulse pressure in the neonatal population. Using a prospective study design in the Regular newborn and Observation nurseries of SIUH, North site. Healthy newborns that are between 0-72 hrs of age will have their blood pressures measured using the oscillometric method. This data will offer insight into whether the presence of wide pulse pressure in otherwise healthy newborn infants warrants further cardiovascular evaluation

ELIGIBILITY:
Inclusion Criteria:

* Infants with gestational age > or = 35weeks and birth weight > 2500g, who are hemodynamically stable, have no cardiorespiratory abnormalities and have no evidence of sepsis. If a blood culture was drawn due to the presence of maternal risk factors (e.g. maternal fever, prolonged rupture of membranes), patients will be included only if the blood culture result is negative and in case of intrapartum antibiotic treatment, ancillary blood tests (CBC with differential, CRP) are also within the normal range

Exclusion Criteria:

* Infants with gestational age < 35weeks or birth weight < 2500g and with evidence of neonatal sepsis either culture proven or clinically suspected.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy newborns in Regular and Observation nurseries who are between 0-72 hrs of age.
Sampling Method: Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
incidence of wide pulse pressures in healthy newborn | 15 mins a day
  This study will determine the incidence of wide pulse pressures in healthy newborn infants during the first days of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

REFERENCES:
- See also: institutional website — http://www.siuh.edu